CLINICAL TRIAL: NCT06032975
Title: Patient-Reported Outcome for Fighting Financial Toxicity in Ovarian Cancer
Brief Title: PRO for Fighting FT in Ovarian Cancer
Acronym: MITO45-ProFFiT
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: MITO 45-ProFFiT
Record Dates: First submitted 2023-08-08; First posted 2023-09-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Financial Toxicity; Quality of life; PROFFIT questionnaire; PRO-CTCAE
MeSH Terms: conditions — Ovarian Neoplasms; Financial Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1:: Patients undergoing their first medical treatment for OC (including adjuvant and neo-adjuvant chemotherapy and first-line treatment for advanced in patients not previously treated with adjuvant chemotherapy)
  Interventions: Other: Questionnaires
- Cohort 2: Patients undergoing their second medical treatment for OC (including the second-line treatment for advanced disease and the first-line treatment for advanced disease in patients previously treated with adjuvant CT)
  Interventions: Other: Questionnaires
- Cohort 3: Patients undergoing their third medical treatment for OC (including the third-line treatment for advanced disease and the second-line treatment for advanced disease in patients previously treated with adjuvant CT)
  Interventions: Other: Questionnaires
- Cohort 4: Patients undergoing their fourth medical treatment for OC (including the fourth- treatment for advanced disease and the third-line treatment for advanced disease in patients previously treated with adjuvant CT)
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The PROFFIT questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where FT can be expressed and is formed by two type of items: (1) outcome (items 1-7) and (2) determinants (items 8-16); EORTC QLQ-C30 questionnaire (items 29-30) and OV28 (items 55-58); PRO-CTCAE: short list of 43 symptoms relevant for ovarian cancer
  Other Names: Questionnaires: PROFFIT, EORTC QLQ-C30 questionnaire (items 29-30), EORTC OV28 (items 55-58), PRO-CTCAE

SUMMARY:
Non-profit, multicenter, prospective, observational study. This study aims to evaluate whether the articulated treatment algorithm that is now possible for OC patients does produce tangible changes of financial distress over the time and whether the determinants of financial distress change their relative weight over the time.

DETAILED DESCRIPTION:
PROFFIT questionnaire is an Italian instrument for evaluating FT in cancer patients in the Italian healthcare context. It includes 16 total items, 7 measuring FT (defining the PROFFIT financial score) and 9 measuring possible determinants of FT.The primary aim of the study is to compare PROFFIT financial score (items 1-7 measuring the financial distress) across different lines of treatment for OC patients undergoing anticancer medical treatment. Primary comparison will be based on PROFFIT questionnaire fulfilled at baseline, before starting each line of treatment.

In addition, among secondary aims of this study, we aim to verify whether FT is associated with quality of life response (items 29-30 of the EORTC QLQ-C30 questionnaire and items 55-56 of the EORTC QLQ-OV28 questionnaire), with patient-self reporting toxicity of treatments (selected symptoms of the PRO-CTCAE library response), and with overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided;
* Women ≥18 years;
* Histologically or citologically confirmed diagnosis of epithelial ovarian, fallopian tube or peritoneal cancer stage IC-IV according to FIGO staging system;
* Patients who are close to begin any type of medical treatment against ovarian cancer.

Exclusion Criteria:

* Major cognitive dysfunction or psychiatric disorders;
* Patients with epithelial ovarian, fallopian tube or peritoneal cancer candidate exclusively to follow-up;
* Patients who have received more than 4 previous lines of medical treatment (maintenance treatments do not represent a line).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Ovarian cancer patients
Study Population: Patients with OC candidate to medical treatment (see cohorts definition).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Financial Toxicity "PROFFIT financial score" | baseline visit, at the end of every cycle of treatment (each cycle is 21 or 28 days depending of type of therapy), and at time of progressive disease (PD) per RECIST 1.1 up to 36 months
  PROFFIT financial score is defined according to items 1-7 of the PROFFIT questionnaire. It will be calculated according to published rules (Riva S, et al. BMJ Open. 2019 Sep;9(9):e031485).

SECONDARY OUTCOMES:
Financial toxicity "Determinants" | baseline visit, at the end of every cycle of treatment (each cycle is 21 or 28 days depending of type of therapy), and at time of progressive disease (PD) per RECIST 1.1 up to 36 months.
  The baseline score for determinants (items 8-16) and their change during treatment
Changes of PROFFIT financial score | baseline visit, at the end of every cycle of treatment (each cycle is 21 or 28 days depending of type of therapy), and at time of progressive disease (PD) per RECIST 1.1 up to 36 months
  Changes of PROFFIT financial score (items 1-7) from baseline during treatment, will be assessed as secondary endpoints.
Quality of Life (QoL) | baseline visit, at the end of every cycle of treatment (each cycle is 21 or 28 days depending of type of therapy), and at time of progressive disease (PD) per RECIST 1.1 up to 36 months
  QoL will be assessed as secondary endpoint using selected QoL items (items 29-30 of the EORTC QLQ-C30 questionnaire, items 55-56 of the EORTC QLQ-OV28 questionnaire) and selected symptoms of the PRO-CTCAE library.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, MD, PhD, Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Nation Cancer Institute of Naples, Division of Medical Oncology - Uro-Gynecology Department, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided